CLINICAL TRIAL: NCT04173858
Title: Evaluation of the Quality of Life of Patients With Opioid-induced Constipation Under Treatment With Naloxegol. A One-year Follow-up Study
Brief Title: Evaluation of the Quality of Life of Patients With Opioid-induced Constipation Under Treatment With Naloxegol
Acronym: KYONAL
Status: Completed | Type: Observational
Sponsor: Kyowa Kirin Farmacéutica S.L.U. (Industry)
Responsible Party: Sponsor
Other Study IDs: KYO-NAL-2017-01
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Opioid-induced Constipation
Keywords: Naloxegol, PAMORA
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Experimental: Patients with confirmed opioid-induced constipation diagnosis and inadequate response to laxatives.
  Interventions: Drug: Naloxegol

INTERVENTIONS:
Drug: Naloxegol — 25 mg oral naloxegol once daily.

SUMMARY:
Opioid-induced constipation (OIC) is a common feature in patients treated with strong opioids. Such medication is often prescribed together with a laxative (osmotic, emollient), with effectiveness depending on the individual patient. Peripherally-acting, mu-opioid receptor antagonists (PAMORAs), such as Naloxegol, have proven to be effective against OIC in patients with inadequate response to laxatives without reducing opioid analgesic effect. However, evidence regarding efficacy and safety on patients with cancer is still scarce. The objective of this study was to analyze the efficacy of naloxegol in a real-world setting by assessing Quality of Life outcomes, and to obtain data on its safety in the long term in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cancer
* Treatment with opioids
* OIC symptoms
* Inadequate response to laxatives
* Karnofsky equal or above 50
* Ambulatory
* Must be able to complete questionnaire forms

Exclusion Criteria: at the start of the study:

* Hypersensitivity to Naloxegol or vehicle
* Suspicion or high risk of gastrointestinal block
* High risk of GI perforation
* Severe liver failure
* Pregnancy or breastfeeding
* Use of potent CYP3A4 inhibitors
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory oncology patients in Spain with diagnosis of OIC.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Assessment of Quality of Life | 12 months
  Patient Assessment of Constipation Quality of Life (PAC-QoL) Questionnaire

SECONDARY OUTCOMES:
Assessment of Constipation Symptoms | 15 days
  Patient Assessment of Constipation Symptoms (PAC-SYM) Questionnaire
Assessment of Constipation Symptoms | 1 month
  Patient Assessment of Constipation Symptoms (PAC-SYM) Questionnaire
Assessment of Constipation Symptoms | 3 months
  Patient Assessment of Constipation Symptoms (PAC-SYM) Questionnaire
Assessment of Constipation Symptoms | 6 months
  Patient Assessment of Constipation Symptoms (PAC-SYM) Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid, Spain